CLINICAL TRIAL: NCT07173348
Title: Effectiveness of Hypnosis on Breathlessness Mastery in Patients With Persistent Dyspnea: a Randomised Controlled Trial
Brief Title: Hypnosis on Breathlessness Mastery in Patients With Persistent Dyspnea
Acronym: HYPNEA
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Geneva (Other)
Collaborators: Lancardis Foundation (Other)
Responsible Party: Principal Investigator, Lisa Hentsch, Head of the outpatient palliative care consultation, University Hospital, Geneva
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2025-00440
Record Dates: First submitted 2025-08-26; First posted 2025-09-15 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Cancer (With or Without Metastasis); COPD III/IV; Interstitial Lung Disease (ILD); Chronic Heart Failure (CHF); Dyspnea
Keywords: Hypnosis; Persistant dyspnea; Cancer with metastasis; Chronic Obstructive Pulmonary Disease; Interstitial Lung Disease; Chronic Heart Failure; Palliative Care
MeSH Terms: conditions — Neoplasms; Lung Diseases, Interstitial; Dyspnea; Pulmonary Disease, Chronic Obstructive | interventions — Hypnosis

STUDY DESIGN:
Intervention Model Description: Open-label, mono-centric, randomised-controlled trial with a two-arm parallel design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hypnosis (Experimental): 3 hypnosis sessions separated by 15 days
  Interventions: Other: Hypnosis
- Usual Care (No Intervention): Usual care

INTERVENTIONS:
Other: Hypnosis — Participants will undergo three 15-minute individual hypnosis intervention, conducted by a trained hypnotherapist, with a two-week interval between each session. A guide for the session has been developed by two experimented hypnotherapists specifically for this intervention and will be used for all sessions. A total of 3 hypnosis session will be realized.
  Arms: Hypnosis

SUMMARY:
Persistent dyspnea is a debilitating symptom, that is common and difficult to treat. This symptom is found in many different diseases including chronic obstructive pulmonary disease (COPD), interstitial lung disease (ILD), chronic heart failure (CHF), and metastatic cancer. Dyspnea is associated with many other symptoms, including anxiety, depression, and fatigue and is responsible for a significant reduction in quality of life. To date, only opiates are recommended for the pharmacological treatment of persistent dyspnea.

The effectiveness of hypnosis is well known in the treatment of anxiety and delivered to patients suffering from chronic dyspnea for this reason. One randomised controlled study has shown that a single 20-minute mindfulness sessions could significantly reduce general symptom burden and have a significant impact on anxiety and depression in palliative care patients. Furthermore, the intervention had no negative side effects.

Our aim is to evaluate the effectiveness of three hypnosis sessions on breathlessness mastery in patients with persistent dyspnea, using as a primary outcome the mastery domain of a validated tool, the Chronic Respiratory Questionnaire (CRQ).

DETAILED DESCRIPTION:
Hypnosis is currently used to reduce anxiety in patients with breathlessness. Although a reduction in anxiety has been correlated with a reduction in dyspnea, the effectiveness of hypnosis on breathlessness self-management has not yet been evaluated. As medical options for the treatment of chronic persistent breathlessness are limited, finding new, innovative ways, to help patients feel more confident in the management of their dyspnea should be a priority. Some interventions such as pulmonary rehabilitation, the hand-held fan and walking aids have been proven to be effective. However, patients with advance disease may not be well enough to endure physical interventions such as pulmonary rehabilitation.

Hypnosis has been shown to be safe and to diminish anxiety in patients suffering from Chronic Obstructive pulmonary disease (COPD). The risk linked to hypnosis is considered minimal as participants may interrupt the hypnosis session at any time and there are no known side effects to hypnosis. Additionally, patients could benefit from the proven reduction of anxiety. The benefits for patients clearly outweigh the risks.

The objective of this prospective parallel randomised controlled trial is to determine the effectiveness of hypnosis on breathlessness mastery in patients with persistant dyspnea and advanced disease. The primary endpoint is the patient-reported breathlessness mastery as measured with the mastery subscale of the Chronic Respiratory Questionnaire (CRQ) after three hypnosis sessions.

Participants will undergo three 15-minute individual hypnosis intervention, conducted by a trained hypnotherapist, with a two-week interval between each session. A guide has been developed by two experimented hypnotherapists specifically for this intervention and will be used for all sessions. The control group will undergo usual care (no hypnosis).

Participants will be recruited at the outpatient consultations of cardiology, pneumology, oncology, primary care and palliative care of the Geneva University Hospital (single centre) by their treating physician. All eligible participants will be presented with the objectives of the study, the procedures involved, the timing of the intervention and will receive an information sheet about the study. Eligible participants will be contacted by a research associate in the following 3 days. If they consent to participate, participants will be randomised to receive either the intervention (3 hypnosis sessions) or usual care.

At inclusion time (T0), all participants will be asked to complete a set of questionnaires: the Chronic Respiratory Questionnaire (CRQ), the Hospital Anxiety and Depression Scale (HADS), the Dyspnea-12 questionnaire (D-12) and the European Quality of Life 5 DImensions 5 Level Version (EQ5D5L), as well as score their worst breathlessness on a numerical scale from 0 to 10, 0 being no breathlessness and 10 worst imaginable breathlessness. These questionnaires will be repeated at the end of the third session. Following the final (third) hypnosis session, participants will be asked about the acceptability of the intervention on a 5-point Likert scale ranging from 0 (not acceptable) to 5 (totally acceptable).

A follow up with the CRQ will be conducted 1 month after the end of the last session.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥ 18 years and
* Primary diagnosis of metastatic cancer, COPD stage at least 3B or E, ILD, or CHF and
* Dyspnea stage NYHA III-IV or mMRC 3-4

Exclusion Criteria:

* Have had hypnosis treatment in the last 12 months
* Have an estimated life expectancy of less than 6 months
* Have participated in pulmonary rehabilitation in the last 6 months
* Have been hospitalised in the last month (30 days)
* Are unable to come to the hospital for 3 outpatient consultations (1 every two weeks)
* Have a condition that would interfere with their ability to respond to the questionnaires (i.e. cognitive impairment, hearing impairment, etc.)
* Are not eligible for a hypnosis session due to a psychiatric disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2027-10-01 (Estimated); Study Completion 2027-10-01 (Estimated)

PRIMARY OUTCOMES:
Chronic Respiratory Questionnaire (CRQ): sub scale mastery | From enrollment to the end of the intervention at 6 weeks.
  The CRQ is a validated 20-item health-related quality of life questionnaire in which experiences are rated on seven-point scales ranging from 1 (maximum impairment) to 7 (no impairment). The CRQ mastery is a domain of the CRQ which comprises four questions with a range of scores also ranging from 1 to 7

SECONDARY OUTCOMES:
Worst breathlessness on the numerical rating scale (NRS) | From enrollment (T0) to the end of the intervention at 6 weeks.
  The numerical rating scale (NRS) ranges from 0 (no breathlessness) to 10 (worst breathlessness).
Physical and affective component of dyspnea with the Dyspnea-12 scale | From enrollment (T0) to the end of the intervention at 6 weeks
  The Dyspnea-12 (D-12) scale is a tool to help to assess the dyspnea. Dyspnea is a multidimensional symptom, comprising physical (intensity, location, temporality and sensory quality) and affective (unpleasant) sensations.
  This D-12 questionnaire is a dyspnea assessment tool. It contains 12 items. The first 7 items correspond to the evaluation of the sensory aspect and the next 5 to the evaluation of the affective aspect. The higher is the score the higher is the burden of dyspnea.
Quality of Life with EQ5D5L | From enrollment (T0) to the end of the intervention at 6 weeks
  The EQ-5D-5L essentially consists of the EQ-5D descriptive system and the EQ visual analogue scale (EQ VAS).
  The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels. The patient is asked to indicate his/her health state by ticking the box next to the most appropriate statement in each of the five dimensions. This decision results in a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state.
  The EQ VAS records the patient's self-rated health on a vertical visual analogue scale where the endpoints are labelled 'The best health you can imagine' and 'The worst health you can imagine'. The VAS can be used as a quantitative measure of health outcome that reflects the patient own judgement.
Acceptability | at the end of the intervention at 6 weeks
  Acceptability will be evaluate at the end of the 3 hypnosis session. with the help of a Lickert scale: completely agree, agree, neutral, don't agree, completely disagree.
Anxiety an Depression (HADS) | From enrollment (T0) to the end of the intervention at 6 weeks
  Anxiety an Depression wil be evaluated with HADS questionnaire which comprises two sub-cathegories, HADS-D for dépression (0-21) and HADS-A for anxiety (0-21)
Duration of hypnosis sessions | After each hypnosis sessions (at 2, 4 and 6 weeks)
  duration in minutes for each hypnosis sessions

OTHER OUTCOMES:
Oxygen saturation | Before and after hypnosis sessions (which will take place at 2,4 and 6 weeks after enrollement).
  Measurement of oxygen saturation through a pulse oximeter in %. It will be measured before and after each session of hypnosis with recording of maximal value
Auto-hypnosis | From enrollment (T0) to the end of the intervention at 6 weeks
  Patient will record the number of auto-hypnosis realized between the sessions of hypnosis in an agenda given at the enrollement in the study.
Heart rate | Before and after hypnosis sessions (which will take place at 2,4 and 6 weeks after enrollement).
  Heart rate ( in beat/min) will be recorded with the help of a pulse oximeter at the finger tip. Maximal value will be recorded after a measurement of 30 seconds.
Respiratory rate | Before and after hypnosis sessions (which will take place at 2,4 and 6 weeks after enrollement).
  Respiratory rate will be recorded counting the number of breathing in 30 seconds and reported in respiration/min.

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Hentsch, Dr med, Principal Investigator — University Hospital, Geneva
Locations (1):
- Geneva University Hospitals, Geneva, Canton of Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: No
No plan to automatically share IPD, but available upon reasonable request once the publication of the study has been made.